CLINICAL TRIAL: NCT03302585
Title: A Phase II Trial of High-Dose Vitamin D Induction in Optic Neuritis (VitaDON 2)
Brief Title: High-Dose Vitamin D Induction in Optic Neuritis
Acronym: VitaDON2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inability to meet recruitment goals
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Jodie Burton MD, MSc, FRCPC, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB17-0922
Record Dates: First submitted 2017-09-27; First posted 2017-10-05 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Optic Neuritis
Keywords: Optic Neuritis; Vitamin D
MeSH Terms: conditions — Optic Neuritis | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: A double-blind randomized placebo/standard therapy phase II trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masked randomization and allocation, only data safety monitor will know allocation if adverse event requires unblinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dose Vitamin D Treatment Group (Experimental): Patients in this arm will receive:
  -5 days of high-dose oral vitamin D3 (50,000 IU daily x 5), followed by 85 days of moderate dose oral vitamin D3 (10,000 IU daily x 85 days)
  Interventions: Drug: Vitamin D3
- Placebo/Standard Vitamin D3 Group (Placebo Comparator): Patients in this arm will receive Placebo/Standard of Care Vitamin D3:
  -5 days of placebo, followed by 85 days of standard of care dose of oral vitamin D3 (4,000 IU daily x 85 days)
  Interventions: Drug: Placebo/Standard of Care Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — 50,000 IU/d of oral vitamin D3 x 5 days followed by 10,000 IU/d of oral vitamin D3 x 85 days
  Other Names: Vitamin D - CHOLECALCIFEROL
  Arms: High-Dose Vitamin D Treatment Group
Drug: Placebo/Standard of Care Vitamin D3 — 50,000 IU/d of oral vitamin D3 x 5 days followed by 40,000 IU/d of oral vitamin D3 x 85 days
  Other Names: Vitamin D - CHOLECALCIFEROL
  Arms: Placebo/Standard Vitamin D3 Group

SUMMARY:
This is a phase II randomized double-blind placebo/standard of care trial to determine if rapidly inducing vitamin D sufficiency in patients with acute optic neuritis results in less damage/greater recovery at 12 months as measured by optical coherence tomography, visual evoked potentials, visual acuity and radiological measures. Our hypothesis, based on earlier observational studies, is that acute optic neuritis in the context of vitamin D sufficiency results in better visual outcomes compared to those that are not sufficient acutely, regardless of such interventions as steroid therapy.

DETAILED DESCRIPTION:
The present trial is based on the observation that vitamin D sufficiency appears to provide some degree of neuroprotection and/or repair in the context of an acute optic neuritis when followed over several months using optical coherence tomography measures. Based on these findings, this randomized double-blinded placebo/standard of care controlled trial has been designed to to see if rapidly inducing vitamin D sufficiency (defined in this trial as a serum 25(OH)D value => 80 nmol/L) results in relatively less reduction in neuroaxonal injury and/or improved recovery chronically (at month 12) versus those patients who do not achieve vitamin D sufficiency in the acute optic neuritis period. of Vitamin D. In this trial, 66 patients in total will be randomized to either "high-dose vitamin D induction" treatment group or the "placebo/followed by standard of care vitamin D" group and followed over 12 months.The primary measure of neuroaxonal integrity in this trial is optical coherence tomography outcomes including ganglion cell layer thickness, retinal nerve fiber layer thickness and macular volume. Other vision metrics and magnetic resonance imaging (MRI) measures will provide secondary outcome indicators of this as well.

ELIGIBILITY:
Inclusion Criteria:

* Canadian residents
* Patients must be between age 18 and 45 years
* Patients must have a diagnosis of either a CIS or RRMS (according to McDonald criteria)
* Patients must have an EDSS of 5.5 or less
* Patients must demonstrate features of a first typical optic neuritis within 21 days of recruitment (or must initiate treatment by day 30)
* Patients must have a baseline 25(OH)D < 80 nmol/L regardless of vitamin D3 supplementation
* Patients must have no contraindications to high-dose vitamin D supplementation
* Female patients must consent to use a reliable form of contraception (oral contraceptive pill, intrauterine device, barrier methods, abstinence) for the duration of the active treatment phase (first 90 days of where study drug provided) of the trial
* Patients must provide written informed consent.

Exclusion Criteria:

* Patients who have had a previous optic neuritis
* Patients with evidence of a non-inflammatory cause of optic neuropathy
* Patients with evidence of neuromyelitis optica spectrum disorder or "NMOSD" (i.e. bilateral optic neuritis, MRI evidence of longitudinally enhancing lesions involving the optic nerves (involving three or more segments of the optic nerve), and/or involving the optic chiasm, and optic tracts
* Patients with a 25(OH)D > 80 nmol/L

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Inter-eye (IED) ganglion cell layer thickness (GCL) | month 12
  The difference between the unaffected and affected eye GCL thickness between treatment and placebo group
Proportion of patients with GCL IED <= 8 microns | 12 months
  The proportion of patients with unaffected and affected eye GCL thickness of < = 8 microns between groups

SECONDARY OUTCOMES:
Change in mean GCL in affected eye over time | baseline to 12 months
  Rate of change in mean GCL thickness in affected eye over study between groups
Change in mean GCL in affected eye over time | baseline to 12 months
  Rate of change in mean GCL thickness in affected eye over study by 25(OH)D level
Change in mean GCL IED between eyes over time | baseline to 12 months
  Rate of change in mean GCL IED thickness in affected eye over study between groups
Change in mean GCL IED between eyes over time | baseline to 12 months
  Rate of change in mean GCL IED thickness in affected eye over study by 25(OH)D level
Change in mean retinal nerve fiber layer (RNFL) in affected eye over time | baseline to 12 months
  Rate of change in mean RNFL thickness in affected eye over study between groups
Change in mean RNFL in affected eye over time | baseline to 12 months
  Rate of change in mean RNFL thickness in affected eye over study by 25(OH)D level
Change in mean RNFL IED between eyes over time | baseline to 12 months
  Rate of change in mean RNFL and GCL thickness in affected eye over study between groups
Change in mean RNFL IED between eyes over time | baseline to 12 months
  Rate of change in mean RNFL and GCL thickness in affected eye over study by 25(OH)D level
Mean RNFL thickness | baseline
  Mean RNFL thickness at baseline and months between groups
Mean RNFL thickness | 1 month
  Mean RNFL thickness at month 1 between groups
Mean RNFL thickness | 6 months
  Mean RNFL thickness at month 6 between groups
Mean RNFL thickness | 12 months
  Mean RNFL thickness at month 12 between groups
Mean GCL thickness | baseline to 12 months
  Mean GCL thickness at baseline between groups
Mean GCL thickness | 1 month
  Mean GCL thickness at month 1 between groups
Mean GCL thickness | 6 months
  Mean GCL thickness at month 6 between groups
Mean GCL thickness | 12 months
  Mean GCL thickness at month 12 between groups
Inter-eye RNFL thickness | baseline to 12 months
  The difference between the unaffected and affected eye RNFL thickness at baseline between treatment and placebo groups
Inter-eye RNFL thickness | 1 months
  The difference between the unaffected and affected eye RNFL thickness at month 1 between treatment and placebo groups
Inter-eye RNFL thickness | 6 months
  The difference between the unaffected and affected eye RNFL thickness at month 6 between treatment and placebo groups
Inter-eye RNFL thickness | 12 months
  The difference between the unaffected and affected eye RNFL thickness at month 12 between treatment and placebo groups
Inter-eye GCL thickness | baseline
  The difference between the unaffected and affected eye GCL thickness at baseline between treatment and placebo groups
Inter-eye GCL thickness | 1 month
  The difference between the unaffected and affected eye GCL thickness at month 1 between treatment and placebo groups
Inter-eye GCL thickness | 6 months
  The difference between the unaffected and affected eye GCL thickness at month 6 between treatment and placebo groups
Inter-eye GCL thickness | 12 months
  The difference between the unaffected and affected eye RNFL thickness between treatment and placebo groups
Mean macular volume (MV) | baseline
  Mean MV at baseline between groups
Mean macular volume (MV) | 1 month
  Mean MV at month 1 between groups
Mean macular volume (MV) | 6 months
  Mean MV at month 6 between groups
Mean macular volume (MV) | 12 months
  Mean MV at month 12 between groups
Mean multifocal VEP (MfVEP) latency | 1 month
  Mean MfVEP at month 1 between groups
Mean change high and low contrast visual acuity (LogMAR) | 12 months
  Mean high and low contrast visual acuity (LogMAR) between groups at from baseline to month 12
Correlation between baseline mean multifocal VEP latency and month-12 GCL, GCL inter-eye difference, RNFL and inter-eye RNFL difference between treatment and placebo groups | 12 months
  Correlation coefficient calculation between mean multifocal VEP latency at baseline and mean GCL, GCL inter-eye difference and RNFL and inter-eye RNFL difference at month 12 between treatment and placebo groups

OTHER OUTCOMES:
Conversion to clinically definite MS (CDMS) | 12 months
  Proportion of patients with clinically isolated syndromes (CIS) who convert to CDMS between groups
New T2 brain lesions on MRI | 12 months
  Mean number of new T2 lesions over study between groups
New contrast enhancing brain lesions on MRI | 12 months
  Mean number of new contrast enhancing lesions over study between groups
Exploratory novel MRI outcomes - diffusion tensor imaging (DTI) | 12 months
  Changes in optic nerve, tract and radiations DTI between groups over study
Exploratory novel MRI outcomes - texture | 12 months
  Changes in optic nerve, tract and radiations texture between groups over study
Exploratory novel MRI outcomes - cross-sectional area | 12 months
  Changes in optic nerve, tract and radiations cross-sectional area between groups over study
Thalamic volume on MRI | 12 months
  Mean thalamic volume over study between groups

CONTACTS AND LOCATIONS:
Overall Officials: Jodie Burton, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No